CLINICAL TRIAL: NCT00816985
Title: Liposuction for Arm Lymphedema Following Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-14728
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: Female; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposuction + Questionnaires (Experimental): Liposuction, followed by Quality of Life Questionnaires and extended follow-up period.
  Interventions: Procedure: Liposuction; Other: Quality of Life Questionnaires

INTERVENTIONS:
Procedure: Liposuction — Liposuction is a procedure that involves the removal of fat from deposits beneath the skin using a hollow stainless steel tube with the assistance of a powerful vacuum. Liposuction can be accomplished either with the use of local or general anesthesia.
Other: Quality of Life Questionnaires — Ratings of 0 to 4, with 0 being Not at ll and 4 being Very Much, regarding how true each statement has been. Statements are in the following categories: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Additional Concerns.

SUMMARY:
The purpose of this study is to determine if a less invasive procedure such as liposuction can be used to effectively reduce arm lymphedema (swelling of the arm) resulting from breast cancer treatment. The standard surgery involves the removal of large portions of skin and tissue leaving a large scar. This less invasive procedure (liposuction) uses 3 to 4 tiny puncture sites and a vacuum tube leaving minimal scars.

ELIGIBILITY:
Inclusion Criteria:

* Patient selection involves identifying women who have undergone breast cancer surgery in the past and who demonstrate lymphedema (stage 2 or 3) based on arm measurement at a minimum of 4 different points along the affected arm. Those women with mild to severe lymphedema with no signs of active infection are candidates for the procedure. History of previous non-surgical treatment for lymphedema will not preclude entry into this trial. All patients must be free of active disease recurrence at study entry. If the lymphedema is of recent onset, then the womans medical oncologist or primary care physician must rule out an underlying cancer recurrence or blood clot.
* Prior therapy including Manuel Lymph Drainage (MLD) or similar massage method, use of compression sleeves, and pneumatic pumps is allowable and may be on-going at study entry. Prior surgical procedures to treat lymphedema such a joining the lymph channels to the blood vessels at any prior time are not eligible for this study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%.
* Life expectancy of greater than one year
* Patients must have normal organ and marrow function as defined below:

  1. leukocytes ≥3,000/MicroL
  2. absolute neutrophil count ≥1,500/MicroL
  3. platelets ≥100,000/MicroL
  4. total bilirubin within normal institutional limits
  5. aspartic transaminase(AST)/alanine transaminase(ALT) ≤2.5 X institutional upper limit of normal
  6. creatinine within normal institutional limits - OR - creatinine clearance ≥60 mL/min/1.73 m² for patients with creatinine levels above institutional normal.
* Able to tolerate general anesthesia and have no recent cardiac history such as myocardial infarction, congestive heart failure, atrial fibrillation, or angina
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents.
* Patients with known metastases should be excluded from this clinical trial because of their poor prognosis.
* History of allergic reactions to compression sleeves, lymphedema bandages, general anesthetics, and all antibiotics
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because: General Anesthesia and/or invasive surgical procedures may increase the risk of miscarriage. Secondly, increased weight during pregnancy may exacerbate lymphedema and thereby make interpretation of the study endpoints difficult.
* Patients with immune deficiency are at increased risk of lethal infections when treated with invasive surgical procedures. Secondly, since this is an elective procedure, the risk to the surgical team of a needle stick would be too high.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-12-03 (Actual); Primary Completion 2011-07-27 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Desired Response | 3 months post last off treatment date
  Investigators plan to show the efficacy of liposuction as a treatment for lymphedema. Investigators will contrast the arm volume at 3 months with the baseline value using a paired t-test. Because the change in volume is likely to be proportional to the baseline value, the logarithm of the volumes will be used. With α = .05 and n = 34, we will have 80% power to detect an effect size of 0.5 (that is, a change of 0.5 standard deviations between the baseline and 3-month mean volumes). However since this is a pilot study with limited funding the study will initially open for 7 patients to assess safety and feasibility.

SECONDARY OUTCOMES:
Number of Participants With Durable Response | Post follow-up period - up to 5 years post treatment
  Durability will be tested for equivalence, by comparing the 3-month and 12-month arm volumes. Five year follow-up is necessary to demonstrate the lasting effect of liposuction in reducing arm lymphedema.
Number of Participants Who Develop an Infection | 12 months per participant
  Measures to reduce skin infections will be implemented in this study but observance of infections will be an important study endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Laronga, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States